CLINICAL TRIAL: NCT01411696
Title: Retrospective Study in Patients Receiving Two or More OZURDEX® Injections for Retinal Vein Occlusion (RVO)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-OZU-09-011; GMA-320 (Other: Allergan, Inc.)
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-03

CONDITIONS: Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Patients who received at least 2 injections of OZURDEX® (dexamethasone intravitreal implant) to treat Macular Edema.
  Interventions: Drug: dexamethasone intravitreal implant 0.7 mg

INTERVENTIONS:
Drug: dexamethasone intravitreal implant 0.7 mg — Dexamethasone intravitreal implant 0.7 mg was dosed previously according to general clinical practice.
  Other Names: OZURDEX®

SUMMARY:
This is a retrospective data collection study to evaluate the efficacy, safety, and re-injection interval of OZURDEX® in the treatment of macular edema due to RVO. Following informed consent, there were no patient study visits. All data was collected via chart review.

ELIGIBILITY:
Inclusion Criteria:

* Macular edema
* Received at least 2 OZURDEX® injections

Exclusion Criteria:

* Received OZURDEX® injections as part of a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received at least 2 injections of OZURDEX® to treat macular edema due to RVO in at least one eye.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Antonio, Texas, United States

REFERENCES:
- [Derived] Dugel PU, Capone A Jr, Singer MA, Dreyer RF, Dodwell DG, Roth DB, Shi R, Walt JG, Scott LC, Hollander DA; SHASTA Study Group. Two or more dexamethasone intravitreal implants in treatment-naive patients with macular edema due to retinal vein occlusion: subgroup analysis of a retrospective chart review study. BMC Ophthalmol. 2015 Sep 4;15:118. doi: 10.1186/s12886-015-0106-z. PMID 26337664
- [Derived] Singer MA, Capone A Jr, Dugel PU, Dreyer RF, Dodwell DG, Roth DB, Shi R, Walt JG, Scott LC, Hollander DA; SHASTA Study Group. Two or more dexamethasone intravitreal implants as monotherapy or in combination therapy for macular edema in retinal vein occlusion: subgroup analysis of a retrospective chart review study. BMC Ophthalmol. 2015 Apr 1;15:33. doi: 10.1186/s12886-015-0018-y. PMID 25885285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 289
Completed | 289
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 289
Age Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 123

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) 4 to 20 Weeks Following the Last OZURDEX® (Dexamethasone Intravitreal Implant) Injection
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). The change in BCVA was calculated using the most improved number of lines read correctly between 4 and 20 weeks following the last injection of OZURDEX® - the number of lines read correctly at baseline. A positive change from baseline indicates improvement.
Time Frame: Baseline, 4 to 20 weeks after last injection (Up to 6 months)
Population: All participants with data available for analysis.
Measure: Mean (Full Range); unit: Lines
Arm/Group | All Participants
Number analyzed (Participants) | 283
Lines
  Baseline | 9.8 (4.62) [0 to 18]
  Change from baseline at Week 4 to 20 (n=209) | 1.0 (3.51) [-13 to 12]

2. Secondary Outcome: Percentage of Participants With an Increase of 2 Lines or More in BCVA
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). An increase of 2 or more lines read correctly compared to baseline is an improvement.
Time Frame: Baseline, Up to 6 months
Population: All participants.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 289
Percentage of participants | 62.9

3. Secondary Outcome: Percentage of Participants With an Increase of 3 Lines or More in BCVA
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). An increase of 3 or more lines read correctly compared to baseline is an improvement.
Time Frame: Baseline, Up to 6 months
Population: All participants.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 289
Percentage of participants | 48.1

4. Secondary Outcome: Change From Baseline in Central Retinal Thickness by Optical Coherence Tomography (OCT) 4 to 20 Weeks After Each Injection
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed in the study eye after pupil dilation at baseline and 4 to 20 weeks after each injection. A negative change from baseline indicates improvement.
Time Frame: Baseline, 4 to 20 Weeks after Each injection (up to 6 months)
Population: All participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: Micron (μm)
Arm/Group | All Participants
Number analyzed (Participants) | 247
Micron (μm)
  Baseline | 437.8 (181.7)
  Change from baseline; first injection (n=242) | -170.8 (179.27)
  Change from baseline; second injection (n=232) | -177.6 (185.21)
  Change from baseline; third injection (n=128) | -160.9 (172.98)
  Change from baseline; fourth injection (n=67) | -155.5 (171.25)
  Change from baseline; fifth injection (n=31) | -145.9 (171.27)
  Change from baseline; sixth injection (n=16) | -193.4 (186.01)
  Change from baseline; seventh injection (n=5) | -220.8 (241.88)
  Change from baseline; eighth injection (n=1) | -75.0 (NA) — No measure of dispersion can be calculated for n=1.
  Change from baseline; ninth injection (n=1) | -61.0 (NA) — No measure of dispersion can be calculated for n=1.

ADVERSE EVENTS:
Description: SAEs (serious adverse events) and AEs (adverse events) were collected retrospectively from chart data.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 7/289
Other Adverse Events (participants affected / at risk) | 49/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=289)
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia (Infections and infestations) | 1
Heart rate irregular (Investigations) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=289)
Cataract (Eye disorders) | 26
Intraocular pressure increased (Investigations) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.